CLINICAL TRIAL: NCT01509430
Title: Progressive Resistance Training as Intervention for Regaining Muscle Mass After Radiation Therapy in Patients With HNSCC - a Randomized Controlled Trial
Brief Title: DAHANCA 25B: Progressive Resistance Training as Intervention for Regaining Muscle Mass After Radiation Therapy in Patients With HNSCC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danish Head and Neck Cancer Group (Network)
Responsible Party: Principal Investigator, Jens Overgaard, Professor, MD, Danish Head and Neck Cancer Group
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: DAHANCA 25B
Record Dates: First submitted 2012-01-03; First posted 2012-01-13 (Estimated); Last update posted 2016-11-29 (Estimated); Status verified 2016-11

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Early training patient (Experimental): 12 weeks of Progressive Resistance Training followed by 12 weeks of a self chosen level of physical activity
  Interventions: Other: Progressive Resistance Exercise Training
- Late training patients (Experimental): 12 weeks of a self chosen level of physical activity followed by 12 weeks of progressive resistance training
  Interventions: Other: Progressive Resistance Exercise Training

INTERVENTIONS:
Other: Progressive Resistance Exercise Training — 12 weeks of Progressive Resistance Exercise Training followed by 12 weeks of self chosen training
  Arms: Early training patient
Other: Progressive Resistance Exercise Training — 12 weeks of self chosen training followed by 12 weeks of progressive resistance exercise training
  Arms: Late training patients

SUMMARY:
Head and neck cancer patients often experience a critical weight loss of around 10% following radiation therapy. Of this up to 70% is muscle mass and is an independent predictor of mortality, lowers muscle strength and functional performance. The purpose of this study is in a randomized controlled trial to investigate the effects of progressive resistance training (PRET) on changes in muscle mass, muscle strength and functional performance in head and neck cancer survivors. The investigators hypothesize that PRET has a positive effect on all primary endpoints and increases muscle mass, muscle strength and functional performance.

ELIGIBILITY:
Inclusion Criteria:

* Histologically diagnosed with squamous cell carcinomas of the larynx (no glottis stage I+II), pharynx, oral cavity or in lymph nodes from an unknown primary tumour (stage I-IV and tumour node metastasis (TNM) classification, UICC, Geneva, 1987)
* Terminated curative radiotherapy treatment with/without chemotherapy;
* No metastases
* Complete tumour remission
* No current or previous malignancies that could prevent participation and training
* No excessive alcohol intake (men > 21 and women > 14 units/wk)
* No recent systematic resistance training or creatine ingestion (within 2 months)
* If woman, not pregnant
* WHO performance status of 0-1
* No psychological, social or geographical conditions that could disturb participation
* Written consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2011-10; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Body composition | Baseline, 3 months and 6 months
  Lean body mass and fat mass assessed by DEXA scanning

SECONDARY OUTCOMES:
Maximal muscle strength | Baseline, 3 months and 6 months
  Isometric and isokinetic muscle dynamometry
Maximal gait speed | Baseline, 3 months and 6 months
  10 m walk time
Patient reported outcomes | Baseline, 3 months and 6 months
  Questionaires on Quality of Life, Fatigue and Mood
Blood sampling | Baseline, 3 months and 6 months
  Investigation of changes in serum level of markers related to weight loss, inflammation and muscle hypertrophy
30 s arm curl capacity | Baseline, 3 months, 6 months
Stair climbing capacity | Baseline, 3 months, 6 months
Jumping capacity | Baseline, 3 months, 6 months
  Counter Movement Jumps
Chair rise capacity | Baseline, 3 months, 6 months
  30 s chair rise

CONTACTS AND LOCATIONS:
Overall Officials: Jens Overgaard, Prof., MD, Principal Investigator — Danish Head and Neck Cancer Group
Locations (1):
- Dept. of Experimental Clinical Oncology, Aarhus C, Denmark

REFERENCES:
- See also: The website for the Danish Head and Neck Cancer Group (DAHANCA). — http://www.dahanca.dk/